CLINICAL TRIAL: NCT07356557
Title: Evaluation of Therapeutic Adherence Among Patients Followed in the Department of Hereditary Metabolic Diseases at Necker Hospital
Acronym: OBSERVANCE MHM
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251413
Record Dates: First submitted 2025-12-17; First posted 2026-01-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Diseases
Keywords: Metabolic disease; Daily oral drug treatment; Medication adherence; Therapeutic education workshop
MeSH Terms: conditions — Metabolic Diseases; Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients, children aged at least 7 years and adolescents/young adults followed in the pediatric department of hereditary metabolic diseases of Necker Hospital, having specific oral drug treatment.
  Interventions: Other: Questionnaire; Other: Calculation of the metabolic balance score

INTERVENTIONS:
Other: Questionnaire — A pseudonymized questionnaire assessing treatment adherence, understanding of the illness, knowledge of medications, and the number of oral medications taken is given to patients and/or their parents during a follow-up visit, whether in a consultation, day hospital, or conventional hospitalization. It is completed by parents and children aged 7 and older, as well as by adolescents and young adults. The responses will not be disclosed to the physicians in the department.
Other: Calculation of the metabolic balance score — For patients with urea cycle deficiency, a metabolic balance score will be calculated independently from retrospective data from the medical record, in the last two years preceding the completion of the questionnaire.

SUMMARY:
The purpose of this study is to evaluate treatment adherence among patients followed in the Department of Inherited Metabolic Diseases at Necker Hospital, in order to assess the need for implementing a therapeutic education workshop focused on medication adherence.

DETAILED DESCRIPTION:
There is limited data in the literature regarding treatment adherence in children with metabolic disorders. A 2011 study on phenylketonuria highlighted a decline in dietary adherence during adolescence. Another study, dating from 1996 and focusing on urea cycle disorders, emphasized the importance of good treatment adherence for maintaining disease control. Furthermore, larger-scale research in epileptic patients has identified several barriers to treatment compliance, highlighting the crucial role of treatment adherence in improving disease control.

The purpose of this study is to evaluate treatment adherence among patients followed in the Department of Inherited Metabolic Diseases at Necker Hospital, in order to assess the need for implementing a therapeutic education workshop focused on medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* All patients followed in the Hereditary Metabolic Diseases department of Necker Hospital during their visit to the department for their usual care and having a specific daily oral medication treatment.
* Children aged at least 7 years and adolescents/young adults
* Holders of parental authority and children or adolescents or adults' patients informed and consenting to participate in the study

Exclusion Criteria:

* Metabolic disease without oral medication (intravenous treatments, amino acid mixtures, and dietary regimens are not evaluated).
* Patient and parents not proficient in French.
* Refusal by the patient's holders of parental authority or adult patient to participate in the study and/or refusal of the child/adolescent.

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients followed in the department of hereditary metabolic diseases at Necker Hospital, having specific oral drug treatment, and having a scheduled care appointment at Necker Hospital as part of their usual follow-up, during the study inclusion period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of therapeutic adherence | Time 0
  Therapeutic adherence score, established from the declarations of patients and their parents to the study questionnaire.

SECONDARY OUTCOMES:
Number of treatments taken each day | Time 0
  Quantification of the number of medications taken daily based on the declarations of patients and their parents to the study questionnaire.
Knowledge of the disease | Time 0
  Assessment of patients' and their parents' knowledge of the disease establish from the declarations of patients and their parents to the study questionnaire.
Knowledge of treatments | Time 0
  Accordance of patients' and their parents' knowledge of treatments, based on the declarations of patients and their parents in the study questionnaire and the patient's prescriptions in the medical record.
Correlation between the therapeutic adherence score and the number of medications taken daily by patients | Time 0
  The therapeutic adherence score and the number of medications taken daily are established from the declarations of patients and their parents to the study questionnaire.
Correlation between the therapeutic adherence score and the age of patients | Time 0
  Therapeutic adherence score, established from the declarations of patients and their parents to the study questionnaire.
Correlation between the therapeutic adherence score and patients' and their parents' knowledge of the disease | Time 0
  The therapeutic adherence score and the knowledge of the disease are established from the declarations of patients and their parents to the study questionnaire.
Correlation between the therapeutic adherence score and patients' and their parents' knowledge of treatments | Time 0
  The therapeutic adherence score and the knowledge of treatments are established from the declarations of patients and their parents to the study questionnaire and on the patient's prescription.
Correlation between therapeutic adherence score and metabolic balance for patients cared for urea cycle deficiency | Time 0
  For patients with urea cycle deficiency, a metabolic balance score will be calculated independently from retrospective data from the medical record, in the last two years preceding the completion of the questionnaire based on the following clinical data:
  * Number of ammonia levels > 100 µmol/L,
  * Mean and median follow-up ammonia levels,
  * Number of glutamine levels > 1000 µmol/L,
  * Number of hospitalizations for decompensation.

CONTACTS AND LOCATIONS:
Overall Officials: Margaux MD GASCHIGNARD, M.D., Principal Investigator — Assistance Publique - Hôpitaux de Paris; Pascale de LONLAY, M.D., PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modi AC, et al. "Adolescent adherence to antiepileptic drug therapy: determinants and clinical outcomes." JAMA, 2011.
- [Background] Maestri NE, et al. "Outcome of urea cycle disorder patients: importance of metabolic control and compliance." Journal of Pediatrics, 1996.
- [Background] Ten Hoedt AE, et al. "Adherence to treatment in phenylketonuria: challenges and improvements." Molecular Genetics and Metabolism, 2011.